CLINICAL TRIAL: NCT07338253
Title: The Effect of the Flipped Learning Model on Spiritual Care Perception and Competence in Nursing Students
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Kağan Arslandoğmuş, Principal Investigator, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KKU-SBE-KA-01
Record Dates: First submitted 2025-12-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Spiritual Care; Flipped Learning Model
Keywords: spiritual care; Flipped Learning Model

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, data will be entered by someone other than the researcher, and statistical analysis will be performed by someone other than the researcher. In the study, the reverse learning model will be applied to participants in the experimental group. As the Flipped Learning Model is an intervention that is clearly noticeable to participants, participants will be aware of which group they are in. This means that blinding participants is not possible. Furthermore, as the researcher is the person implementing the intervention, both participants and the researcher will be aware of the intervention. Therefore, blinding will not be performed in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flipped Learning Model (Experimental): Receiving Spiritual Care Training in Nursing with the Reverse Education Model
  Interventions: Other: flipped learning model
- TRADITIONAL EDUCATION MODEL (No Intervention): Receiving spiritual care training in nursing with the traditional education model

INTERVENTIONS:
Other: flipped learning model — All participating students will be administered the 'Introductory Characteristics Form', the 'Spirituality and Spiritual Care Rating Scale (MMBÖ)' and the 'Spiritual Care Competence Scale (MBYÖ)' and a pre-test. Students in the experimental group will undergo reverse application for one month.
  All students in the control group will be administered the 'Descriptive Characteristics Form,' the 'Spirituality and Spiritual Care Rating Scale (MMBÖ),' the 'Spiritual Care Competence Scale (MBYÖ),' and the pre-test. No intervention will be administered to students in the control group.
  After the reverse application is completed, the 'Descriptive Characteristics Form', the 'Spirituality and Spiritual Care Rating Scale (MMBÖ)' and the 'Spiritual Care Competence Scale (MBYÖ)' and the 'post-test' will be administered to the students in the experimental and control groups.
  Arms: Flipped Learning Model

SUMMARY:
The Effect of the Flipped Learning Model on Nursing Students' Perception of Spiritual Care and Competence This study was designed as a randomised controlled trial to determine the effect of the flipped learning model on nursing students' perception of spiritual care and their competence in spiritual care.

The study will be conducted between 08.12.2025 and 09.02.2026 on 112 fourth-year nursing students. Students meeting the inclusion criteria will be randomised and divided into two random groups: the experimental group (n=50) and the control group (n=50). All participating students will be administered the 'Descriptive Characteristics Form', the 'Spirituality and Spiritual Care Rating Scale (MMBÖ)' and the 'Spirituality Scale Spiritual Care Competence Scale (MBYÖ)' and (pre-test). Students in the experimental group will undergo reverse application for 1 month.

All students in the control group will be administered the 'Descriptive Characteristics Form,' the 'Spirituality and Spiritual Care Rating Scale (MMBÖ),' the 'Spiritual Care Competence Scale (MBYÖ),' and a pre-test. No intervention will be administered to students in the control group.

After the reverse application is completed, the 'Descriptive Characteristics Form,' the 'Spirituality and Spiritual Care Rating Scale (MMBÖ),' the 'Spiritual Care Competence Scale (MBYÖ),' and the 'post-test' will be administered to the students in the experimental and control groups.

The collected data will be analysed using SPSS 22 software.

ELIGIBILITY:
Inclusion Criteria:

* Students who volunteer to participate in the study, who have smartphones/computers and continuous Internet access, will be included in the study.

Exclusion Criteria:

* Students who have previously studied a health-related subject and who have previously taken a course related to spiritual care will be excluded from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2025-12-28 (Actual); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Determining the effect of the flipped learning model on nursing students' perception level of spiritual care | Baseline and post-intervention (8th week)]
  Spirituality and Spiritual Care Rating Scale (SCRS); The scale consists of 17 items and has 3 sub-dimensions. The scale is scored using a 5-point Likert type (1 = Strongly Disagree, 2 = Disagree, 3 = Undecided, 4 = Agree, 5 = Strongly Agree). Thirteen items (1, 2, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, and 17) are scored normally, while four items (3, 4, 13, and 16) are scored in reverse. The total score is obtained by dividing the item scores by the number of questions. The maximum score that can be obtained from the scale is 85, and the minimum is 17. A high total score indicates a good level of perception of spirituality and spiritual care concepts.
  The Spiritual Care Competence Scale (SCCS) consists of three areas of nursing competence related to spiritual care and a total of 27 items. The scale is a five-point Likert-type scale. The lowest possible score on the scale is 27, and the highest possible score is 135. A high score indicates nursing competence related to spiritual care.

SECONDARY OUTCOMES:
Determining the effect of the flipped learning model on nursing students' their spiritual care competencies | Baseline and post-intervention (8th week)]
  Spirituality and Spiritual Care Rating Scale (SCRS); The scale consists of 17 items and has 3 sub-dimensions. The scale is scored using a 5-point Likert type (1 = Strongly Disagree, 2 = Disagree, 3 = Undecided, 4 = Agree, 5 = Strongly Agree). Thirteen items (1, 2, 5, 6, 7, 8, 9, 10, 11, 12, 14, 15, and 17) are scored normally, while four items (3, 4, 13, and 16) are scored in reverse. The total score is obtained by dividing the item scores by the number of questions. The maximum score that can be obtained from the scale is 85, and the minimum is 17. A high total score indicates a good level of perception of spirituality and spiritual care concepts.
  The Spiritual Care Competence Scale (SCCS) consists of three areas of nursing competence related to spiritual care and a total of 27 items. The scale is a five-point Likert-type scale. The lowest possible score on the scale is 27, and the highest possible score is 135. A high score indicates nursing competence related to spiritual care.

CONTACTS AND LOCATIONS:
Overall Officials: Kağan ARSLANDOĞMUŞ, Principal Investigator — Kırıkkale University
Locations (1):
- Kirikkale University, Kırıkkale, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No